CLINICAL TRIAL: NCT05666544
Title: Developing and Effectiveness Evaluation of Web-based Situation Renal Replacement Therapies Patient Decision Aids
Brief Title: Renal Replacement Therapies Decision Aids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUH109-REC3-085
Record Dates: First submitted 2022-12-06; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: End-stage Renal Disease; Renal Replacement Therapy; Decision Aid; Decision-making
Keywords: End-stage Renal Disease; Renal Replacement Therapy; Patient Decision Aid; Shared Decision-Making
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written health education leaflets (Active Comparator): Using written health education leaflets to conduct education.
  Interventions: Other: Written health education leaflets
- Web-based patient decision aid (Experimental): Using web-based patient decision aid of renal replacement therapy.
  Interventions: Other: Web-based patient decision aid

INTERVENTIONS:
Other: Web-based patient decision aid — After the clinic, use web-based patient decision aid of renal replacement therapy to conduct education.
  Arms: Web-based patient decision aid
Other: Written health education leaflets — After the clinic, use a written health education leaflet on renal replacement therapy to conduct education.
  Arms: Written health education leaflets

SUMMARY:
Different renal replacement therapy methods will cause significant impacts on the physical, mental, and social for patients with end-stage renal disease. Application shared decision-making should be able to effectively assist patients in choosing suitable renal replacement therapy. Currently, most of the patient decision aid of renal replacement therapy are written health education leaflets, which have problems such as too many words, more difficult content, and inconvenience. In shared decision-making, even though different treatment options are communicated to patients, there is still a gap between "understanding" and "real experience", it will be creating uncertainty of decision, and emphasizing true situational learning strategies should be a viable auxiliary method. Therefore, this study aims to develop a web-based patient decision aid of renal replacement therapy and integrates situational learning strategies into it. First, investigators have conducted a qualitative study to explore the related experience of patients with end-stage renal disease the decision-making needs in renal replacement therapy choice, and the experience and barrier of reading paper patient decision aid. Next, based on the results of the pilot study, the modified Delphi method will be used to collect the opinions of experts, and the situational learning theory will be integrated into the patient decision aid to develop the web-based situation renal replacement therapies patient decision aid. After completion, investigators will apply quasi-experimental, a repeated measurement that will be adopted to analyze the effectiveness of web-based patient decision aid of renal replacement therapy in shared decision-making in patients with end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by nephrologists as patients with chronic kidney disease, and GFR <30 ml/min/1.73m2.
* As a patient admitted to the "Pre-ESRD care plan".
* Clear awareness, ability to communicate in Mandarin and Taiwanese, and agree to participate in the research.
* Those who are unable to answer the questions without other serious diseases or diseases affecting the mind.

Exclusion Criteria:

* Those who cannot freely choose hemodialysis or peritoneal dialysis due to absolute contraindications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes to the Preparation for Decision Making Scale (PrepDMS) | Baseline and immediately post-intervention.
  The PrepDMS is a self-reported instrument assessing perceptions of usefulness in communicating health decisions. Possible scores range from 1(not at all) to 5 (a great deal). The higher the score, the higher the readiness for decision-making.
Changes to the Decisional Conflict Scale (DCS) | Baseline, immediately post-intervention, and one-month post-intervention.
  The DCS is a self-reported instrument assessing individual conflict and uncertainty about decision-making. Possible scores range from 0 (strongly agree) to 4 (strongly disagree). The higher the score, the higher the decisional conflict.
Changes to the Decision Self Efficacy Scale (DSES) | Baseline, immediately post-intervention, and one-month post-intervention.
  The DSES is a self-reported instrument assessing an individual's confidence or belief in their ability to make decisions. Possible scores range from 0 (not at all conflict) to 4 (very conflict). The higher the score, the higher the decision-making self-efficacy.
Decision Regret Scale (DRS) | One-month post-intervention.
  The DRS is a self-reported instrument measuring regret about health-related decisions. Possible scores range from 1 (strongly agree) to 5 (strongly disagree). Higher scores indicate higher decision-making regret.
Changes to the Renal Replacement Therapy Knowledge Scale (RRTKS) | Baseline and immediately post-intervention
  The RRTKS is a self-reported instrument to assess knowledge of different treatment modalities. Scored as correct (1 point) and incorrect (0 points). Higher scores indicate higher knowledge of different treatment modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis JL, Davison SN. Hard choices, better outcomes: a review of shared decision-making and patient decision aids around dialysis initiation and conservative kidney management. Curr Opin Nephrol Hypertens. 2017 May;26(3):205-213. doi: 10.1097/MNH.0000000000000321. PMID 28212179
- [Background] Gionfriddo MR, Leppin AL, Brito JP, Leblanc A, Boehmer KR, Morris MA, Erwin PJ, Prokop LJ, Zeballos-Palacios CL, Malaga G, Miranda JJ, McLeod HM, Rodriguez-Gutierrez R, Huang R, Morey-Vargas OL, Murad MH, Montori VM. A systematic review of shared decision making interventions in chronic conditions: a review protocol. Syst Rev. 2014 Apr 15;3:38. doi: 10.1186/2046-4053-3-38. PMID 24731616
- [Result] Bailey RA, Pfeifer M, Shillington AC, Harshaw Q, Funnell MM, VanWingen J, Col N. Effect of a patient decision aid (PDA) for type 2 diabetes on knowledge, decisional self-efficacy, and decisional conflict. BMC Health Serv Res. 2016 Jan 14;16:10. doi: 10.1186/s12913-016-1262-4. PMID 26762150
- [Result] Buhse S, Muhlhauser I, Heller T, Kuniss N, Muller UA, Kasper J, Lehmann T, Lenz M. Informed shared decision-making programme on the prevention of myocardial infarction in type 2 diabetes: a randomised controlled trial. BMJ Open. 2015 Nov 13;5(11):e009116. doi: 10.1136/bmjopen-2015-009116. PMID 26567256
- [Derived] Su JM, Kuo HL, Yang KL, Wu CJ, Ho YF. Interactive decision aid on therapy decision making for patients with chronic kidney disease: A prospective exploratory pilot study. Digit Health. 2025 Apr 1;11:20552076251332832. doi: 10.1177/20552076251332832. eCollection 2025 Jan-Dec. PMID 40177120